CLINICAL TRIAL: NCT03714997
Title: Mechanisms and Efficacy of High-intensity Training in Motor Incomplete Spinal Cord Injury
Brief Title: High Intensity Exercise in Incomplete SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Rehabilitation Hospital of Indiana (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, George Hornby, Professor of Physical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1806265450; CDMRP-eBRAP-SCI170299 (Other Grant/Funding Number: Department of Defense - Clinical Trials)
Record Dates: First submitted 2018-07-25; First posted 2018-10-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Parallel design randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded outcomes assessment at each measures phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Locomotor Training (Experimental): High Intensity Locomotor Training will consist of 30 sessions of walking related activities in variable contexts (i..e, on a treadmill, overground, and on stairs), with a primary goal to achieve 40 minutes of walking within 1 hour sessions while achieving heart rates close to 80% of heart rate reserve.
  Interventions: Procedure: Walking training
- Low Intensity Locomotor Training (Active Comparator): High Intensity Locomotor Training will consist of 30 sessions of walking related activities in variable contexts (i..e, on a treadmill, overground, and on stairs), with a primary goal to achieve 40 minutes of walking within 1 hour sessions while achieving heart rates from 30% to 40% of heart rate reserve.
  Interventions: Procedure: Walking training

INTERVENTIONS:
Procedure: Walking training — Practice of walking training in variable contexts, including multiple tasks and environments specific to the patients' deficits and community walking goals.
  Other Names: Locomotor training; Walking Exercise; Gait Training

SUMMARY:
The goal of this study is to identify the comparative efficacy of high-intensity walking training in individuals with chronic, motor incomplete spinal cord injury as compared to lower-intensity walking exercise.

DETAILED DESCRIPTION:
Background/Readiness: The objective of this proposal is to maximize locomotor outcomes of patients following incomplete spinal cord injury (iSCI) through identification of rehabilitation strategies that maximize recovery. Specific training parameters, such as provision of large amounts of stepping, appears to facilitate locomotor function in patients with iSCI, although other factors may be critical. In this proposed phase II randomized clinical trial, the overarching hypothesis is that the "intensity" of locomotor practice, defined as power output and estimated using cardiopulmonary measures, is critical to maximizing walking outcomes. Performance of high intensity locomotor training increases the cardiovascular and neuromuscular demands, which results in physiological changes that facilitate greater locomotor performance in individuals with and without neurological injury. There are, however, limited data supporting its utility in patients with iSCI. Recent findings suggest a role for high-intensity stepping training in variable contexts, with gains in peak locomotor capacity as compared low-intensity variable training. Additional changes in cardiopulmonary function and neuromuscular coordination provide a mechanistic rationale for the utility of this strategy. Such changes are likely due to increased central (volitional) activation, and are in sharp contrast to the long-standing notion that high intensity training impairs motor function in neurological injury.

Despite these data, genotypic variations suggest specific caveats related to high intensity training. For example, many patients possess a single nucleotide polymorphism (SNP) variation in the brain derived neurotrophic factor (BDNF) gene that may impact the activity-dependent BDNF expression thought to contribute to neuroplasticity underlying improved performance. This single nucleotide polymorphism (SNP) can influential declarative memory, with recent data suggesting a potential impact on motor recovery after neurologic injury. Previous studies indicate limited BDNF increases in patients with this SNP during high intensity exercise, although the effects of locomotor recovery with repeated high-intensity training is unclear Hypothesis/Specific Aims: The primary hypotheses are that high intensity variable stepping can markedly improve locomotor performance as well as neuromuscular and cardiopulmonary function as compared to lower-intensity training in patients with chronic motor iSCI. It is believed that genotypic variations in the ability to synthesis activity dependent BDNF may modify the effects of high intensity training. Specific Aim 1: Test if high intensity stepping training in variable contexts results in greater locomotor gains as compared to lower intensity interventions. Specific Aim 2: Test the effects of these training strategies on neuromuscular and cardiopulmonary impairments. Specific Aim 3: Test the effects of the presence of the BDNF SNP on locomotor improvements in patients following high-intensity activities Study Design: This phase II, stratified, assessor- blinded randomized clinical trial will assess the effects 2 months (up to 30 sessions) of high- vs low-intensity variable stepping training on ambulatory patients with chronic (> 1year) motor iSCI. Participants referred from outpatient therapy settings will undergo evaluation of locomotor performance, cardiopulmonary capacity, and neuromuscular coordination and impairments prior to and following each training paradigm, with 2-month follow-up assessments.

Clinical Impact: The application of high-intensity locomotor training in the clinical rehabilitation of patients with iSCI is extremely limited, despite data regarding the potential benefits in neurological intact individuals and patients with stroke. The clinical application of high-intensity training represents a simple, readily modified training parameter that can be readily implemented, and is in stark contrast to current clinical practice and challenge traditional dogma in rehabilitation medicine.

ELIGIBILITY:
Inclusion criteria

* Individuals with motor incomplete SCI (AIS C or D) > 12 mo. duration will be recruited to participate in the study, with further criteria including anatomical lesions between C1-T10..
* Participants will be between 18 and 75 years of age (note: while participants > 50 yrs with subacute SCI have a reduced probability of functional ambulation 79, participants will already be ambulatory with only minimal or no assistance and in the chronic phase of rehabilitation, and prediction rules using age will not necessarily apply in this study).
* All participants must be able to perform walking training with passive range of motion within the limits of normal locomotor function, including: 0-30 degrees ankle plantarflexion, knee flexion from 0 to 90 degrees, hip flexion to 0-90 degrees.

Exclusion criteria:

* Participants with body mass > 400 lbs will be excluded, which is the highest limit for use of our motorized treadmill and safety harness systems.
* Participants will be medically stable with medical clearance to participate, with absence of concurrent severe medical illness including: unhealed decubiti, existing infection, significant cardiovascular or metabolic disease which limits exercise participation, significant osteoporosis (as indicated by history of fractures following injury), active heterotrophic ossification in the lower extremities, known history of peripheral nerve injury in lower legs, history of traumatic brain injury, and history of pulmonary complications that limits exercise capacity, including significant obstructive and/or restrictive lung diseases.
* Participants who are ventilator-dependent will be excluded secondary to severely impaired respiratory capacity.
* Participants with substantial orthopedic bracing to stabilize the cervical or thoracic vertebral column are not eligible due to safety concerns with harness supported ambulation training..
* Patients will also be excluded if they are unable to tolerate 10 minutes of standing without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic); previous experience in the sub-acute population suggests that 10 minutes of standing is more than sufficient for tolerating 45 minutes of walking secondary to increased activity/muscle pump minimizing risk for orthostasis.
* Individuals who are undergoing concurrent physical therapy will be excluded from the study population to eliminate confounding effects of additional physical interventions, Other therapies, such as occupational or speech therapies, will be allowed as prescribed by their physician. Individuals will be allowed and encouraged to continue their normal exercise routines during the course of the intervention, with activity monitors measuring stepping activity in all participants
* Women of childbearing potential will not be excluded, although women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion.
* All subjects prescribed oral anti-spastic medications will not be excluded, although patients with intrathecal baclofen pumps or history of recent (< 3 months) botulinum toxin injection in the lower extremities will be excluded due to potential increases in weakness interfering with the effects of stepping training performance.
* Patients with a known history of autonomic dysreflexia will not be excluded, although specific signs and symptoms of all patients with history of injury > T6 anatomical level will be closely monitored throughout training.

Other criteria

* Men and women will be recruited for participation in the proposed clinical trial at rates consistent with national and local average of gender disparities of SCI (80% male, 20% women). Women of childbearing potential will not be excluded, although women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion.
* Individuals of different ethnicities will be recruited at rates similar to the national and local ethnicity rates. Current data since 2005 indicate that of the entire population of SCI, 66.1% are Caucasian, 27.1% are African American, 6.6% are of Hispanic origin, and 2.0% Asian. These populations closely resemble those at RHI and in our previous studies in human SCI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Fastest overground walking speed | Changes from baseline to post-testing at 8 weeks
  fastest walking speed during 10 m walk test
peak treadmill speed | Changes from baseline to post-testing at 8 weeks
  fastest treadmill speed reached for 1 full minute on graded exercise test

SECONDARY OUTCOMES:
6 min walk test | Changes from baseline to post-testing at 8 weeks
  distance walked over 6 min
self-selected speed | Changes from baseline to post-testing at 8 weeks
  self-selected speed during 10 m walk test

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Hornby TG, Plawecki A, Lotter J, Shoger L, Voigtmann C, Heffron L, Lucas E, Parrott D, Henderson CE. Higher Intensity Walking Training in Individuals With Chronic Motor Incomplete Spinal Cord Injury: A Randomized Clinical Trial. Neurorehabil Neural Repair. 2026 Jan;40(1):49-60. doi: 10.1177/15459683251399158. Epub 2025 Dec 27. PMID 41454653